CLINICAL TRIAL: NCT05854901
Title: Procalcitonin-guided Treatment Regarding Antibiotic Use for Acute COPD Exacerbations: a Prospective Randomised Controlled Trial
Brief Title: PCT-guided Treatment Regarding Antibiotic Use for Acute COPD Exacerbations
Acronym: PRECISION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Menno M. van der Eerden, Principal investigator and Pulmonologist, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NL72662.078.20; NL9122 (Registry Identifier: Netherlands Trial Register)
Record Dates: First submitted 2023-02-14; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: COPD Exacerbation; COPD; Acute Copd Exacerbation
Keywords: Procalcitonin
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized clinical multi-center study to evaluate procalcitonin-guided treatment regarding antibiotic use in patients who are admitted because of an acute COPD exacerbation. Patients who are admitted are randomly assigned to either procalcitonin-guided treatment (in which antibiotics are started when the procalcitonin concentration is above 0.25 ng/mL) or usual care in which the treating physician decides whether or not to start with antibiotic treatment. Patients will be stratified for study center.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCT-guided treatment (Experimental): Patients randomized to this arm will only receive antibiotic treatment when the procalcitonin concentration is > 0.25ug/L.
  Interventions: Diagnostic Test: Procalcitonin
- Usual care (Active Comparator): Patients randomized to this arm will receive antibiotic treatment based on the physician's decision.
  Interventions: Other: Physician's decision

INTERVENTIONS:
Diagnostic Test: Procalcitonin — blood test, measuring the concentration of PCT in ug/L
  Other Names: PCT
  Arms: PCT-guided treatment
Other: Physician's decision — The physician's decided whether the patient will receive antibiotic treatment or not
  Arms: Usual care

SUMMARY:
This study the investigators will examine whether procalcitonin-guided treatment regarding antibiotic therapy is non-inferior to usual care in patients who are admitted because of an acute COPD exacerbation when it comes to treatment failure on day 30.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a prevalent disease, worldwide, and in the Netherlands with approximately 600.000 patients. COPD is currently the 3rd leading cause of death worldwide and is also a leading cause of disability-adjusted life years. Given the contribution of exacerbations both to loss in quality of life and to health-care costs, it is of paramount importance to improve the current treatment of exacerbations.

Pulmonary physicians are well aware of overuse of antibiotics, but lack the tools to decide which medication to give in the clinical setting. Biomarkers may aid towards a more personalized treatment of acute COPD exacerbations (AECOPD). Procalcitonin (PCT), the precursor of calcitonin, is released in response to a bacterial infection by many tissues within 6-12 hours after the onset of infection, while the concentration is only minimally raised in viral infections, making it a relative specific diagnostic tool for bacterial infection. Several trials have shown a reduction in antibiotic consumption in AECOPD when using a PCT-guided treatment algorithm. Recent systematic reviews concluded that appropriately powered trials are lacking to confirm that clinical outcomes are comparable with usual care.

In this study the investigators will examine whether a PCT-guided treatment regarding antibiotic therapy is non-inferior to usual care in patients who are admitted because of an acute COPD exacerbation when it comes to treatment failure on day 30.

ELIGIBILITY:
Inclusion Criteria:

* COPD, according to GOLD 2018 definition
* Indication for hospitalization because of acute severe exacerbation of COPD, as defined by GOLD 2018 and modified Anthonisen criteria
* Presence of at least 2 major symptoms of the modified Anthonisen criteria (acute deterioration in sputum volume, sputum purulence and dyspnea) or the presence of 1 major symptom and 1 minor symptom (coughing, wheeze, nasal discharge, sore throat, fever)
* Post-bronchodilator FEV1/FVC < 0,70 and FEV1% < 80%pred. within last 5 years
* At least 40 years
* Smokers or ex-smokers with > 10 packyears
* Written informed consent
* Start of symptoms no more than 7 days before admission

Exclusion Criteria:

* Indication for ICU and or non-invasive ventilation < 72h of admission
* Pneumonia, radiologically confirmed
* Infection at another site and/or sepsis according to the SIRS criteria (with tachycardia and tachypnea not being caused by the exacerbation)
* COPD before age 40
* Asthma, without presence of COPD.

  * Patients with COPD , with or without a history of asthma (in childhood or as an adolescent) will NOT be excluded/are allowed to participate.
  * Patients with Asthma/COPD overlap syndrome (with current asthma AND COPD) will NOT be excluded/are allowed to participate.
* Clinically relevant heart failure or myocardial ischemia
* Chronic use of immunosuppressants, including prednisolone (a prednisone equivalent of 10mg or less is allowed/is NOT an exclusion criterion)
* Known bronchiectasis as a primary diagnosis
* Colonisation with Pseudomonas spp. or other micro-organisms in recent cultures (last 60 days) not susceptible to amoxicillin-clavulanic acid
* Pregnancy
* Recent exacerbation (last 28 days)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 693 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | 30 days
  Treatment failure is defined as disease-related mortality, need for endotracheal intubation or vasopressors, renal failure (defined as Kidney Disease: Improving Global Outcomes (KDIGO) stage 3 - new renal replacement therapy, tripling of baseline creatinine, or serum creatinine > or = 350 umol/L), lung abcess/empyema, development of pneumonia or rehospitalization within 30 days after inclusion.

SECONDARY OUTCOMES:
Incomplete resolution of the clinical signs and symptoms | change between baseline and after 30 days
  Incomplete resolution of the clinical signs and symptoms associated with the AECOPD at day 30 after inclusion of the study (i.e. not reaching the baseline condition prior to the AECOPD) scored using the modified Anthonisen criteria
Incomplete resolution of the clinical signs and symptoms | day 30
  Incomplete resolution of the clinical signs and symptoms associated with the AECOPD at day 30 after inclusion of the study (i.e. not reaching the baseline condition prior to the AECOPD) scored using the modified Anthonisen criteria
Modified Anthonisen criteria | baseline
  Patients fill in the modified Anthonisen criteria card on day 1 as a baseline measure
Modified Anthonisen criteria | day 3
  Patients fill in the modified Anthonisen criteria card on day 3
Modified Anthonisen criteria | day 5
  Patients fill in the modified Anthonisen criteria card on day 1 as a baseline measure
Modified Anthonisen criteria | day 10
  Patients fill in the modified Anthonisen criteria card on day 1 as a baseline measure
Decision to start antibiotic therapy after an initial opposite decision (after 48 hours) | 30 days
  Decision to start antibiotic therapy after an initial opposite decision (after 48 hours)
Side effects of antibiotic treatment | 30 days
  Side effects of antibiotic treatment, such as gastro-intestinal complaints, allergic reactions
Cumulative antibiotic consumption | 30 days
  The cumulative amount of antibiotic treatment consumed by the patient during follow-up
Cumulative prednisolone consumption | 30 days
  The cumulative amount of prednisolone consumed by the patient during follow-up
Length of hospitalization | up to 30 days
  Duration of time (in days) of the admission in hospital for the index exacerbation during follow-up
Re-exacerbation | 30 days
  The presence of a new exacerbation, requiring treatment (prednisolone and/or antibiotic treatment) during follow-up
EXACT respiratory questionnaire | change between baseline and after 30 days
  PROM symptom score: EXACT - Respiratory symptoms scale
EXACT respiratory questionnaire | baseline
  PROM symptom score: EXACT - Respiratory symptoms scale
EXACT respiratory questionnaire | day 10
  PROM symptom score: EXACT - Respiratory symptoms scale
EXACT respiratory questionnaire | day 30
  PROM symptom score: EXACT - Respiratory symptoms scale
CAT | baseline
  COPD assessment test, quality of life questionnaire
CAT | day 10
  COPD assessment test, quality of life questionnaire
CAT | day 30
  COPD assessment test, quality of life questionnaire
CAT | change between baseline and day 30
  COPD assessment test, quality of life questionnaire
EQ-5D-5L | baseline
  quality of life questionnaire
EQ-5D-5L | day 10
  quality of life questionnaire
EQ-5D-5L | day 30
  quality of life questionnaire
EQ-5D-5L | change between baseline and day 30
  quality of life questionnaire
iMCQ | 30 days
  Medical consumption questionnaire, measuring the total amount of medical consumption (admission, ER visits, outpatient visits) during follow-up
Non-invasive ventilation after 72 hours of admission | 30 days
  Need for non-invasive ventilation after 72 hours of admission
Time to complete resoluation of symptoms | 30 days
  · Time to complete resolution of symptoms according to daily symptom diaries evaluating the modified Anthonisen criteria

OTHER OUTCOMES:
Cost-effective analysis | 30 days
  Alongside the clinical trial, an economic evaluation will be performed conform the guidelines of the Health Care Institute Netherlands (17). This evaluation will be conducted from a societal and payer's perspective. When adopting the societal perspective, costs will include 30-day inpatient and outpatient (emergency room, specialist visits) hospital costs, primary care costs (visits to GP and nurse practitioner), medication costs, ambulance costs, productivity costs, informal care costs and travel costs.

CONTACTS AND LOCATIONS:
Overall Officials: Menno M van der Eerden, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (11):
- Netherlands (11):
  - Zuyderland hospital, Heerlen, Limburg
  - Amphia hospital, Breda, North Brabant
  - Catharina hospital, Eindhoven, North Brabant
  - Bravis hospital, Roosendaal, North Brabant
  - Noordwest hospital group, Alkmaar, North Holland
  - OLVG, Amsterdam, North Holland
  - MST Enschede, Enschede, Overijssel
  - Isala klinieken, Zwolle, Overijssel
  - Groene Hart, Gouda, South Holland
  - Erasmus MC, Rotterdam, South Holland
  - Franciscus Gasthuis & Vlietland, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Netherlands Trial Register registration included in ICTRP — https://trialsearch.who.int/Trial2.aspx?TrialID=NL9122

DOCUMENTS (2):
  • Study Protocol (2022-08-23): https://cdn.clinicaltrials.gov/large-docs/01/NCT05854901/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/01/NCT05854901/SAP_001.pdf